CLINICAL TRIAL: NCT06285786
Title: Does Proper Patient Handling Technique, Coupled With New Technology, Help Reduce Musculoskeletal Demands of Health Care Workers
Brief Title: Patient Handling Techniques and New Technology for Health Care Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of New Brunswick (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REB 2023-109
Record Dates: First submitted 2023-10-13; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-12

CONDITIONS: Work-related Injury
Keywords: Patient Handling; Injury Prevention; Technology; Intervention; Training

STUDY DESIGN:
Intervention Model Description: One single group of participants will be performing the same patient handling tasks:
  1. During session 1 (Pre-Intervention) participants will not receive any instruction on how to perform the patient handling techniques on both beds.
  2. During session 2 (Post-Intervention) participants will be asked to perform the patient handling techniques as seen during the intervention on both beds.
Masking Description: Participants will be masked of the proper technique/training during the pre-intervention session (with and without the use of technology). Specifically, on how to manually move the patient in both beds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing Student (Experimental): The study involves 1 single arm. A single group of participants will experience all experimental conditions. From an ergonomic standpoint, it has been recognized that providing patient-handling ergonomics training is crucial to their safety. This project will compare the same group performing patient handling tasks without training versus training while utilizing both long term care beds.
  Interventions: Other: Ergonomic Training on Patient Handling Techniques

INTERVENTIONS:
Other: Ergonomic Training on Patient Handling Techniques — Each participant will receive an ergonomic training on proper patient handling technique, adhering to the appropriate program to use with the SAMS bed and the Vendlet between session 1 & 2.
  In small groups of 6-10 participants, a healthcare ergonomist (M. Leger) will be responsible to demonstrate, instruct and evaluate each participant on all 4 techniques on the SAMS bed. Each participant will have multiple opportunities to demonstrate their skills.
  In the same session, each participant will also receive proper training from a specialized occupational therapist on how to use the Vendlet. Each participant will have multiple opportunities to demonstrate their skills.
  After completing the intervention, each participant will be prepared to participate in the post-intervention data collection session in the laboratory.

SUMMARY:
Patient handling is a major risk-factor for the development of musculoskeletal injuries in healthcare providers. To have a significant impact on injury reduction related to patient handling will require the incorporation of technology. This project is to investigate a piece of technology that has been designed to facilitate in-bed patient handling: The Vendlet.

The purpose of this research project is to assess the ability of the Vendlet system outfitted on a Span-America Medical Systems (SAMS) bed to reduce the physical load on healthcare providers performing patient handling tasks. This evidence-based outcomes will be used to support the mitigation of the Vendlet from the European market into the Canadian market. The SAMS bed is currently available in North America and has several adjustable features to support patient transfer activities.

The project will provide a biomechanical comparison of commonly used patient handling techniques performed using a SAMS bed outfitted with and without a Vendlet patient transfer device. This Vendlet technology has the potential to significantly reduce the musculoskeletal and joint strain of healthcare providers while handling patients.

DETAILED DESCRIPTION:
The General Objectives of this project are as followed:

1. The first research objective is to build complex movement waveform models to help assess kinematic, neuromuscular and force demands related to patient handling and the associated human movement patterns. These waveform models will then be used to best answer our two main research questions.
2. The second research objective is to build a biomechanical shoulder and back model to determine the cumulative load (joint stresses) demands related to patient handling as a means to quantify the risk of injury at these highly vulnerable joints. These cumulative loading models will then be used to best answer our two main research questions.
3. The third and last research objective is to determine the margin of error of a markerless motion capture system compared to a gold standard marker-based motion capture system; to determine the feasibility for future research to be conducted in a health care setting and thus increasing the ecological validity of the assessment during a typical working day.

This project has the following Research Questions:

1. What are the movement technique patterns and physical demands associated with performing patient handling techniques with and without the use of medical bed assistive technology?
2. What effect does training have on patient handling techniques? Specifically, does training help improve the healthcare worker's movement patterns as well as reduce physical load demands?

This project has the following Research hypotheses:

1. It is hypothesized that the use of technology (Vendlet system coupled with the SAMS bed) will reduce the physical demands of healthcare providers while handling patients.
2. Training safe patient handling techniques will result in safer patient handling practices and reduce physical demands while handling patients due to improved movement techniques.

Introduction

This project will provide a biomechanical comparison of commonly used patient handling techniques, performed using a Span-America Medical Systems (SAMS) long-term care bed outfitted with and without a Vendlet patient turning system. The Vendlet is a powered patient turning aid that replaces the bed-rail system of the hospital bed. Using a set of rollers that can be adjusted for height, the Vendlet mechanically moves the bed sheet beneath the patient in a controlled manner. The system can assist in turning the patient, as well as repositioning them in the bed. The SAMS long-term care bed is highly adjustable, has been designed to facilitate patient handling and was designed around patient safety. The researchers will investigate both technologies (the Vendlet and SAMS long-term care bed) and quantify the reduction physical demands of patient handling when combined.

Methods:

30 nursing students will be recruited from a regional university and college programs. Diversity in participant recruitment will be based on the enrolment proportion in the regional postsecondary programs. Each participant will be required to attend two different sessions:

1. During the first session, participants will receive full instructions on how to use the SAMS Advantage Ready Wide bed and the Vendlet system and will be provided with time to familiarize themselves with the technology. Participants will perform 4 different patient repositioning techniques associated with turning the patient: 1- reposition the patient vertically to the head of the bed. 2- repositioning horizontally in bed from one side to the other side of the bed. 3- turning a patient from their back to their side, away from the caregiver. 4- placing the patient in a sling. Each of the techniques will be performed with the two medical bed configurations: a) the SAMS Advantage Ready Wide hospital bed on its own; and b) with the Vendlet system mounted on the SAMS bed. The order of the repositioning techniques will be randomized, and each patient repositioning technique will be performed 3 times.

   Once the first session is completed, each participant will receive the intervention: proper training on patient handling care, as well as proper training on technology use, while handling a patient by a healthcare ergonomist (M. Léger) and an occupational therapist (P. Beck).
2. During the second session, participants will return to the laboratory to perform the same 4 different patient repositioning techniques, using both bed configurations, while applying their new training techniques.

Throughout all experimental sessions, the following equipment will be used: 1- Motion capture system (to track individual motions and patient handling performances and develop a biomechanical model to assess joint stress); 2- Surface electromyography (EMG) (to monitor neuromuscular activity and effort); 3- galvanic skin response system and a heart rate monitor (to assess levels of stress); 4- Pressure Mats (bed and foot mats will be used to measure pressure distribution/load demands of handling a patient. Participants' feedback will also be recorded using exit surveys.

Statistical Analysis

A factorial repeated measure mixed analysis of variance (ANOVA) with a within factors (independent variables: techniques) and two between factor (beds and training) will be performed to evaluate differences between movement patterns, neuromuscular activity, perceived discomfort, heart rate, electrodermal activity, foot pressure distribution and bed pressure distribution (dependent variables). Prior to running the factorial repeated measures ANOVA, Skewness and Kutosis will be assessed for normal distribution with a z-score set at 3,29. The Mulchy's test will be used to assess the sphericity assumption. When the sphericity assumption is violated, the Greenhouse Geiser will be used as a correction. The Alpha level will be set at p < .05, and if any significant interactions are found, the Tukey correction will be used as a post hoc analysis. Principal Component Analysis will be incorporated to determine the modes of variation in both the kinematic and kinetic (shoulder and joint loads) biomechanical motion patterns (waveforms), while performing the patient handling techniques with and without the incorporated technology.

ELIGIBILITY:
Inclusion Criteria:

- One-month history of no pain or injury in the low back or shoulder region.

Exclusion Criteria:

- Participant received a training on proper patient handling techniques.

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular Activity - Average muscle activation | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Eight bilateral muscles will be examined: anterior deltoid [AD], trapezius descendens [TD], biceps brachii [BB], thoracic erector spinae [TES] located at the level of the T9 spinous process, lumbar erector spinae [LES] located at the level of the L3 spinous process, external oblique [EO], rectus femoris [RF], and biceps femoris [BF]. The raw EMG signal will be rectified, and Butterworth low passed filtered (RMS converted) using MATLAB. Peak activity will be found for each muscle during the maximum voluntary contraction (MVC) trials and used to normalize all subsequent EMG data. Therefore, the EMG data will represent a percent change from the participants' MVCs for each muscle, during each patient handling trial. An analysis of the neuromuscular activation changes (%MVC) will be compared during each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Neuromuscular Activity - Peak muscle activation | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Eight bilateral muscles will be examined: anterior deltoid [AD], trapezius descendens [TD], biceps brachii [BB], thoracic erector spinae [TES] located at the level of the T9 spinous process, lumbar erector spinae [LES] located at the level of the L3 spinous process, external oblique [EO], rectus femoris [RF], and biceps femoris [BF]. The raw EMG signal will be rectified, and Butterworth low passed filtered (RMS converted) using MATLAB. Peak activity will be found for each muscle during the maximum voluntary contraction (MVC) trials and used to normalize all subsequent EMG data. Therefore, the EMG data will represent a percent change from the participants' MVCs for each muscle, during each patient handling trial. An analysis of the neuromuscular activation changes (%MVC) will be compared during each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Motion Capture: To assess postural changes in patient handling technique. | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Kinematic coordinates of markers will be gap filled (spline smoothing algorithm) and then filtered using a 2nd order Butterworth low pass filter (cut off frequency of 10Hz). Visual 3D, C-motion software will be used to filter raw kinematic data as well as calculate specific joint angles. 3D movement (flexion/extension, lateral bend, and twist) of the neck, both arms, pelvis, trunk-pelvis, hips, knees, and trunk-thigh will be used in Visual 3D to calculate three-axis joint angles. Visual 3D software will be used to calculate kinematic and kinetic values. The kinematics (joint angles) and kinetics (inverse dynamics) will be compared for each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Motion Capture: To assess cumulative load forces | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Kinematic coordinates of markers will be gap filled (spline smoothing algorithm) and then filtered using a 2nd order Butterworth low pass filter (cut off frequency of 10Hz). Visual 3D, C-motion software will be used to filter raw kinematic data as well as calculate specific joint angles. 3D movement (flexion/extension, lateral bend, and twist) of the neck, both arms, pelvis, trunk-pelvis, hips, knees, and trunk-thigh will be used in Visual 3D to calculate three-axis joint angles. Visual 3D software will be used to calculate kinematic and kinetic values. Visual 3D will also be used to calculate the inverse dynamics of the participants; calculating kinetics will help us determine the force and cumulative load demands of the participant while they handle a patient. The kinematics (joint angles) and kinetics (inverse dynamics) will be compared for each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Motion Capture: To assess joint angles | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Kinematic coordinates of markers will be gap filled (spline smoothing algorithm) and then filtered using a 2nd order Butterworth low pass filter (cut off frequency of 10Hz). Visual 3D, C-motion software will be used to filter raw kinematic data as well as calculate specific joint angles. 3D movement (flexion/extension, lateral bend, and twist) of the neck, both arms, pelvis, trunk-pelvis, hips, knees, and trunk-thigh will be used in Visual 3D to calculate three-axis joint angles. Visual 3D software will be used to calculate kinematic and kinetic values. The kinematics (joint angles) and kinetics (inverse dynamics) will be compared for each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Foot Pressure Distribution: Peak pressure will be the outcome measure of interest to assess postural balance and stability of the participant performing the patient handling technique. | Post-intervention (within 2 weeks after intervention)
  The Xsensor FOOT and GAIT software (Xsensor, Calgary, AB, Canada) will be used to measure the peak pressure in each section of the patient's sole and plantar contact area during each patient handling techniques. To study the pressure variations in greater detail, the foot data will be subdivided into the following : 1- the toe (T); 2- the metatarsals (M) separated into three parts (metatarsal 1: M1, metatarsal 2&3: M2, metatarsal 4&5: M3); 3- the midfoot (MF); and 4- the heel (H) separated into two parts (medial heel: MH, and lateral heel: LH) . Peak pressure values will also be assessed for each section of the foot during each patient handling techniques. The foot pressure distribution outcomes will be compared between each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Foot Pressure Distribution: Contact area will be the outcome measure of interest to assess postural balance and stability of the participant performing the patient handling technique. | Post-intervention (within 2 weeks after intervention)
  The Xsensor FOOT and GAIT software (Xsensor, Calgary, AB, Canada) will be used to measure the peak pressure in each section of the patient's sole and plantar contact area during each patient handling techniques. To study the pressure variations in greater detail, the foot data will be subdivided into the following : 1- the toe (T); 2- the metatarsals (M) separated into three parts (metatarsal 1: M1, metatarsal 2&3: M2, metatarsal 4&5: M3); 3- the midfoot (MF); and 4- the heel (H) separated into two parts (medial heel: MH, and lateral heel: LH). Peak pressure values will also be assessed for each section of the foot during each patient handling techniques. The foot pressure distribution outcomes will be compared between each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Bed Pressure Distribution: Average pressure distribution will be outcome measures to assess the safe placement of the patient. | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Bed Pressure Distribution will be considered in four body regions at two-time points on both beds. The body regions include the right and left regions of the back (including the shoulders and upper back) and the right and left areas of the pelvis (hips). These regions will be compared at two separate time points: the initial participant position (lying supine prior to any patient handling technique) and the final participant position (once the patient handling technique is completed). At each timepoint, pressure-related outcome measures will be computed for each task. Contact area (in2), average pressure on contact area (mmHg), and peak pressure will be among the outcome measures (mmHg). The bed pressure distribution outcomes will be compared between each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.
Bed Pressure Distribution: Peak pressure distribution will be outcome measures to assess the safe placement of the patient. | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Bed Pressure Distribution will be considered in four body regions at two-time points on both beds. The body regions include the right and left regions of the back (including the shoulders and upper back) and the right and left areas of the pelvis (hips). These regions will be compared at two separate time points: the initial participant position (lying supine prior to any patient handling technique) and the final participant position (once the patient handling technique is completed). At each timepoint, pressure-related outcome measures will be computed for each task. Contact area (in2), average pressure on contact area (mmHg), and peak pressure will be among the outcome measures (mmHg). The bed pressure distribution outcomes will be compared between each patient handling technique between 1- SAMS bed (with the Vendlet) vs the SAMS bed (without the Vendlet), and 2- Pre vs Post Intervention.

SECONDARY OUTCOMES:
Self Reported Questionnaires | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  Rate of Perceived Discomfort (RPD) questionnaire used to quantify participants perceived discomfort while performing a patient handling technique. The RPD is a self-reported questionnaire with a 100-point visual analogue scale that indicates the level of discomfort relative to specific body parts.
Exit Survey | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  At the end of each patient handling techniques (with and without the Vendlet) a second questionnaire will be used to quantify bed preference, by asking the participants: Which bed did you prefer while performing the patient handling technique?
Rating of Perceived Exertion (RPE) | Pre-Intervention and Post-intervention (within 2 weeks after intervention)
  The Rating of Perceived Exertion (RPE) questionnaire is a modified Borg Scale to quantify effort (CSEP-SCPE, 2023). The modified Borg Scale is a 0-10 scale where 0 correspond to "Very Light Activity", and 10 correspond to "Maximum Effort".

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Wayne J Albert, PhD., Doctorate, Principal Investigator — University of New Brunswick; Dre. Michelle Cardoso, PhD, Doctorate, Principal Investigator — Universite de Moncton
Locations (1):
- Universite de Moncton, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang Y, Wang D, Ying J, Chu P, Qian Y, Chen W. Design and Preliminary Validation of Individual Customized Insole for Adults with Flexible Flatfeet Based on the Plantar Pressure Redistribution. Sensors (Basel). 2021 Mar 4;21(5):1780. doi: 10.3390/s21051780. PMID 33806449
- [Background] Budarick AR, Moore C, Fischer SL. Evaluating patient turn effectiveness using turn-assist technologies. J Med Eng Technol. 2020 Jan;44(1):1-11. doi: 10.1080/03091902.2019.1707889. Epub 2020 Jan 15. PMID 31939691